CLINICAL TRIAL: NCT06195410
Title: The Effect of Mother and Father Kangaroo Care on Newborn and Parent Outcomes in Premature Infants: A Randomized Cross Over Study
Brief Title: The Effect of Mother and Father Kangaroo Care on Newborn and Parent Outcomes in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SelcukU-12c-2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Kangaroo Care
Keywords: Mother Kangaroo Care; Father Kangaroo Care; Cross Over Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator: Intervention Group (Active Comparator)
  Interventions: Other: kangaroo care application
- Comparator (Sham Comparator)
  Interventions: Other: kangaroo care application

INTERVENTIONS:
Other: kangaroo care application — In the study, the mother applied kangaroo care to her premature baby for 65 minutes, and after a 24-72 hour washout period, the father applied kangaroo care for 65 minutes.

SUMMARY:
First aim is to determine the effect of mother and father kangaroo care on the premature baby's Comfort Behavior level and physiological parameters (respiratory rate, heart rate, oxygen saturation and body temperature). Second aim is to determine the effect of mother and father kangaroo care on Parental Satisfaction and Neonatal Intensive Care Parental Stress level.

The study was a a randomized crossover study with pretest-posttest design. It was carried out in the neonatal intensive care unit of Selçuk University Faculty of Medicine Hospital in Konya province. Study data were collected from 19 mother and 19 father and their premature newborns between February 2023 and August 2023.

DETAILED DESCRIPTION:
In the study, the mother applied kangaroo care to her premature baby for 65 minutes, and after a 24-72 hour washout period, the father applied kangaroo care for 65 minutes. The order of mother and father application was determined randomly.

Data were collected using Physiological Parameters Form, Neonatal Comfort Behavior Scale, Parental Satisfaction Scale and Neonatal Intensive Care Unit Parental Stress Scale.

In the study, physiological parameters and Neonatal Comfort Behavior Scale scores of premature infants and Neonatal Intensive Care Unit Parental Stress Scale and Parental Satisfaction Scale scores of parents were evaluated. Pearson Chi-Square Test, Yates Correction and Fisher's Exact Test were used to compare categorical data according to groups. Two Independent Sample t Test was used to compare normally distributed variables and Mann Whitney U Test was used to compare non-normally distributed variables. Statistical significance level was accepted as p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

For premature infants;

* The baby is born before 36+6 weeks of gestation Stability of vital parameters at the time of application, Stable health status (cardiorespiratory stability, no congenital or chromosomal abnormalities, no history of intraventricular hemorrhage, no history of periventricular leukomalacia and NEC, no systemic and metabolic disorders),

For parents;

* Willingness to participate in the research
* Being able to read and write Turkish

Exclusion Criteria:

For premature infants;

* Being connected to a mechanical ventilator
* Congenital or chromosomal abnormality
* Being with deprivation syndrome
* Having a history of intraventricular hemorrhage

For parents:

* Not being willing to care for kangaroos
* Having a physical disability to care for kangaroos

Ages: 26 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Physiological parameters of the premature infant:respiration rate | Change from baseline, 30min, and 65 min
  The infant's is respiratory rate per minute.
Physiological parameters of the premature infant:peak heart rate | Change from baseline, 30min, and 65 min
  The infant's is heart rate per minute. Philips IntelliVue MP40 device was used to monitor heart rete.
Physiological parameters of the premature infant: oxygen saturation | Change from baseline, 30min, and 65 min
  Oxygen saturation measures the percentage of oxyhemoglobin (oxygen-bound hemoglobin) in the blood, and it is represented as arterial oxygen saturation (SaO2) and venous oxygen saturation (SvO2). Philips IntelliVue MP40 device was used to monitor %SpO2.
Physiological parameters of the premature infant: body temperature | Change from baseline, 30min, and 65 min
  Shows body temperature.
Comfort Behavior scale scores of the premature infant | Change from baseline, 30min, and 65 min
  Comfort Behavior scale was used. The Neonatal Comfort Behavior Scale (NEAS) is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. Each item in the scale is scored from 1 to 5. It is evaluated over the total score. The lowest score that can be obtained from the Newborn Comfort Behavior Scale (NEAS) is 6, and the highest score is 30.
Parent Satisfaction points | baseline and 70 min
  Parental Satisfaction scale was used. This scale was developed to assess parents' satisfaction in NICU. EMPATHIC-30 scale, 1= definitely not; 6 = absolutely yes and consists of five sub-dimensions; information (5 items), care and treatment (8 items), organization (5 items), parent involvement (6 items) and the professional attitude of the staff (6 items). One point represents the lowest satisfaction, while 6 points represents the highest satisfaction.
Neonatal Intensive Care Unit Parental Stress Scale points | baseline and 70 min
  Neonatal Intensive Care Unit Parental Stress Scale was used.The scale is a 34-item Likert-type scale with three subscales (Sights and Sounds, Infant Behavior and Appearance, and Parental Role Changes). Responses to the scale rate parents' stress level for each item from 1 (not at all stressful) to 5 (very stressful). As the scale score increases, stress increases.

CONTACTS AND LOCATIONS:
Overall Officials: Busra Yahsi, Principal Investigator — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No